CLINICAL TRIAL: NCT02303873
Title: Efficacy and Safety of Alendronate in Chinese Children or Adolescents With Osteogenesis Imperfecta: an Age Stratified Prospective Study
Brief Title: Efficacy and Safety of Alendronate in Chinese Children or Adolescents With Osteogenesis Imperfecta
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No. 2007-03-12
Record Dates: First submitted 2014-11-19; First posted 2014-12-01 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-11

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Alendronate

ARMS (1):
- an open label, prospective, self-controlled study (Experimental): Children or adolescents under the age of 18 years old with minor trauma fracture were recruited from 30 provinces of China. The diagnosis of OI was made by endocrinology department of Peking Union Medical College Hospital(PUMCH).
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Alendronate — Alendronate was administrated as 70 mg/week orally (Fosamax, Merck Sharp & Dohme．LTD.).

SUMMARY:
Alendronate should be considered as an alternative therapy of osteogenesis imperfecta (OI) because it significantly increased areal bone mineral density (BMD) and its Z score, decreased fracture incidence, inhibited bone resorption biomarkers. Alendronate exerted beneficial roles in different age brackets, especially in young patients with OI.

ELIGIBILITY:
Inclusion Criteria:

1. children or adolescents aged 0-18 years,
2. had either a history of at least once minor-impact fracture or age and sex adjusted areal BMD Z score of -1.0 or less at lumbar spine or total hip;
3. with or without blue sclera, impaired hearing, joint hypermobility or dentinogenesis imperfecta;
4. with or without slim long bone; with or without cranial epactal bones, signs of multiple fractures, bony deformity in skeletal X-ray films.

Exclusion Criteria:

1. previous history of rickets, hyperparathyroidism, other metabolic or inherited bone diseases; malignant disease; coeliac disease; hyperthyroidism;
2. therapy history of BPs within recent two years; severe renal failure (creatinine clearance <40 ml/min), chronic liver disease; severe diseases of gastrointestinal tract;
3. unable to keep upright for at least 30 minutes daily .

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2007-03; Primary Completion 2011-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
changes from baseline of areal BMD at lumbar spine and total hip | baseline and 12,24,36 months
annual clinical fracture incidence | baseline and 12,24,36 months

SECONDARY OUTCOMES:
changes of bone turnover biomarkers | baseline and 6,12,24,36 months
changes of height | baseline and 12,24,36 months